CLINICAL TRIAL: NCT02042950
Title: A Phase II Study of Carfilzomib in the Treatment of Relapsed/Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0259; NCI-2014-01271 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Mantle Cell Lymphoma; MCL; Relapsed; Refractory; Carfilzomib
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Recurrence | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib given at a dose of 20*/56 mg/m^2 (* CFZ 20 mg/m2 by vein on Days 1 and 2 in Cycle 1 followed by 56 mg/m^2 for each subsequent dose thereafter) on days 1 and 2, 8 and 9, 15 and 16 of a 28-day cycle (following cycle 12 carfilzomib given on days 1 and 2 and 15 and 16 only).
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Starting dose: 20 mg/m2 by vein on Days 1 and 2 in Cycle 1 followed by 56 mg/m^2 for each subsequent dose thereafter) on days 1 and 2, 8 and 9, 15 and 16 of a 28-day cycle (following cycle 12 carfilzomib given on days 1 and 2 and 15 and 16 only).

SUMMARY:
The goal of this clinical research study is to learn if carfilzomib can help control relapsed or refractory MCL. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If participant is found to be eligible for this study, they will begin the first cycle of treatment with carfilzomib. Each cycle is 28 days.

On Days 1, 2, 8, 9, 15, and 16 of Cycles 1-12:

* Participant will receive carfilzomib by vein over 30 minutes. The first 2 doses participant receives may be lower than later doses. This is to reduce the risk of an allergic reaction.

On Days 1, 2, 15, and 16 of Cycles 13 and beyond:

* Participant will receive carfilzomib by vein over 30 minutes.

Participant should drink at least 6-8 cups (8 ounces each) of fluid per day starting 2 days before their first day of treatment and for as long as their doctor asks them to. During Cycles 1 and 2, participant will receive fluids by vein before and after their dose of carfilzomib.

Before participant receives carfilzomib, they will be given standard drugs (such as allopurinol, dexamethasone, antibiotics, anti-fungals, and/or anti-virals) to help decrease the risk of side effects. Participant may ask the study staff for information about how the drugs are given and their risks.

When participant receives the drugs during Cycle 1 and on Day 1 of Cycle 2, they will be monitored for side effects for 1 hour after they receive the study drug.

Study Visits:

On Day 1 of all cycles:

* Participant will have a physical exam.
* Participant will have a neurological exam to check for weakness, numbness and pain in their hands and feet.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If participant's doctor thinks it is needed, they will have a bone marrow biopsy and/or aspiration to check the status of the disease.
* If participant's doctor thinks it is needed, they will have an ECHO or a MUGA.
* If participant is able to become pregnant, they will have a blood (about 1½ tablespoons) or urine pregnancy test. (Cycles 2 and beyond only)

On Days 2, 9, and 16 of all cycles:

* Participant's vital signs will be measured.

On Days 8 and 15 of all cycles:

* Participant will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If participant is able to become pregnant, they will have a blood (about 1½ tablespoons) or urine pregnancy test.

On Day 1 of Cycles 2, 4, 6, and so on up to Cycle 12, then every 3 cycles after that:

* If the study doctor thinks it is needed, participant will have a CT scan, MRI, PET scan, and/or PET/CT scan to check the status of the disease.
* If the study doctor thinks it is needed, participant will have a gastrointestinal endoscopy or colonoscopy.

Length of Study:

Participant may continue taking the study drug for up to 3 years. Participant will no longer be able to take the drug if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over once they have completed the long term follow-up phone calls.

End-of-Treatment Visit:

Within about 30 days, after participant finishes taking the study drug they will return to the clinic for the following tests and procedures:

* Participant will have a physical exam.
* Participant will have a neurological exam to check for weakness, numbness and pain in their hands and feet.
* Participant will have an EKG to check their heart function.
* Blood (about 3-5 tablespoons) will be drawn for routine tests and to check the status of the disease.
* Participant will have a CT scan and/or x-ray to check the status of the disease.
* Participant will have a PET/CT scan to check the status of the disease.
* If participant's doctor thinks it is needed, they will have a bone marrow biopsy and aspiration
* If participant's doctor thinks it is needed, they will have a colonoscopy/gastrointestinal endoscopy.
* If participant is able to become pregnant, they will have a blood (about 1½ tablespoons) or urine pregnancy test.

Long Term Follow-Up:

After participant's end-of-treatment visit, they will be called every 6 months for 1 year to see how they are doing and to find out about any other treatments they have received since they stopped study treatment. These calls will take about 2-3 minutes. In addition to the phone calls, participant's medical records may be reviewed as well.

This is an investigational study. Carfilzomib is FDA approved and commercially available for the treatment of certain types of multiple myeloma. This drug is investigational for the treatment of MCL.

Up to 60 participants will be enrolled on this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of mantle cell lymphoma.
2. Patients must have relapsed or refractory MCL.
3. Understand and voluntarily sign an IRB-approved informed consent form.
4. Age >/= 18 years at the time of signing the informed consent.
5. Patients must have bi-dimensional measurable disease (bone marrow only involvement is acceptable).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
7. Serum bilirubin <1.5 mg/dl and Creatinine Clearance >/= 30 mL/min, platelet count >50,000/mm^3 and absolute neutrophil count (ANC) > 1,000/mm^3. [Patients who have bone marrow infiltration by MCL are eligible if their ANC is ≥ 500/mm^3 (growth factor allowed) or their platelet level is equal to or > than 30,000/mm^3.]. AST (SGOT) and ALT (SGPT) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present. Uric acid within normal limits.
8. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test within 30 days of initiation of therapy. * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
9. FCBP must agree to use a highly-effective form of birth control while taking the study drug and for 1 month after the last dose of study drug. Highly-effective forms of birth control include implants, injectables, birth control pills with 2 hormones, some intrauterine devices (IUDs), or having a sterilized partner. The type of birth control used must be discussed with and approved by the attending physician prior to initiation of study drug.
10. Males must agree to use a condom with spermicide every time they have sex during the study and for 3 months after the last dose of study drug. They also must agree to not donate sperm during the study and for 3 months after the last dose of study drug.
11. Patients must be willing to receive transfusions of blood products.

Exclusion Criteria:

1. Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active hemorrhage, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Known HIV infection. Patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation
4. All patients with active central nervous system lymphoma.
5. Significant neuropathy (Grades 3 - 4, or Grade 2 with pain) within 14 days prior to enrollment.
6. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
7. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis to ascites requiring paracentesis.
8. Patients with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment).
9. Patients with symptomatic bradycardia (heart rate < 50 bpm, hypotension, light-headedness, syncope).
10. Use of any standard/experimental anti-lymphoma drug therapy, including steroids, within 3 weeks of initiation of the study or use of any experimental non-drug therapy (e.g. donor leukocyte/mononuclear cell infusions) within 56 days of initiation of the study drug treatment. Prior allogeneic SCT within 16 weeks or autologous SCT within 8 weeks of initiation of therapy.
11. Patients with New York Health Association (NYHA) Class III and IV heart failure, myocardial infarction in the preceding 6 months, and conduction abnormalities, including but not limited to atrial fibrillation, atrioventricular (AV) block block, QT prolongation, sick sinus syndrome, ventricular tachycardia, as these patients may be at greater risk for cardiac complication, per carfilzomib labeling.
12. The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent. Investigator discretion is allowed.
13. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment.
14. Patients who have received any previous Carfilzomib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07-14 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hun J. Lee, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 6 enrolled participants 2 failed screening.
Groups:
- Carfilzomib: To evaluate the efficacy of single agent carfilzomib in patients with relapsed/refractory MCL as measured by response rate.
Period: Overall Study
Arm/Group | Carfilzomib
Started | 4
Completed | 0
Not Completed | 4
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Carfilzomib
Description: To evaluate the efficacy of single agent carfilzomib in patients with relapsed/refractory MCL as measured by response rate.
Time Frame: 21 months
Population: Unable to complete final analysis due to not meeting enrollment requirements.
Arm/Group | Carfilzomib
Number analyzed (Participants) | 0

2. Other Pre Specified Outcome: Toxicity of Carfilzomib
Description: To further evaluate the toxicity of Carfilzomib in patients
Time Frame: 21 months
Population: Unable to complete final analysis due to not meeting enrollment requirements.
Arm/Group | Carfilzomib
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Post Treatment
Description: To estimate the response duration, progression free survival, time to failure and overall survival.
Time Frame: 21 months
Population: Unable to complete final analysis due to not meeting enrollment requirements.
Arm/Group | Carfilzomib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | Carfilzomib
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=4)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=4)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Alk Phos Increase (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (5)
AST Increase (Investigations) | 1 (1)
Bili Rubin Increase (Investigations) | 1 (1)
Blurred Vision (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine Increase (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3)
Dry Eyes (Eye disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema Limbs (General disorders) | 1 (1)
Elevated BUN (Metabolism and nutrition disorders) | 3 (4)
Elevated Lactic Acids (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 4 (7)
Fever (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperhidrosis (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesium (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil Decrease (Investigations) | 1 (3)
Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Platelet Count Decrease (Investigations) | 4 (9)
White Blood Cell Decrease (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT02042950/Prot_SAP_000.pdf